CLINICAL TRIAL: NCT06003868
Title: Investigation of the Effect of Hippotherapy Simulator on Balance and Walking in Children With Spastic Diplegia Cerebral Palsy
Brief Title: Investigation of the Effect of Hippotherapy Simulator in Children With Spastic Diplegia and Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, assistant professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar72
Record Dates: First submitted 2023-08-11; First posted 2023-08-22 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy; Balance; Distorted; Walking, Difficulty
Keywords: Cerebral palsy; hippotherapy; walking; balance; life quality; diplegia
MeSH Terms: conditions — Cerebral Palsy; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Exercises with Hippotherapy Simulator: This exercise will be applied to the group for 8 weeks, 2 days a week, as a single session (15 minutes) a day. The patients will be placed on the simulator and the starting position will be taught. They will be warned to maintain the starting position throughout the movements of the simulator. The hippotherapy simulator will be operated almost in the gait pattern of the horse and in the 1st stage of the 3-stage speed level. If the patients have unusual complaints such as dizziness, blackout, chest pain and risk of falling during the application. they will be advised to request to stop the application
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Physiotherapy will be applied for 8 weeks, 2 days a week, as one session per day (45 minutes).
  Interventions: Other: traditional physiotherapy
- hippotherapy group (Experimental): Physiotherapy will be applied for 8 weeks, 2 days a week, one session a day (45 minutes). In addition, the patients will be placed on the simulator and the starting position will be taught. your simulator They will be warned before and during the application to maintain the starting position throughout their movements.
  pattern and will be run in the 1st stage of the 3-stage speed level.
  Interventions: Other: traditional physiotherapy; Other: hippotherapy-assisted physiotherapy

INTERVENTIONS:
Other: traditional physiotherapy — Stretching for patients with spasticity exercises walking exercises for balance and gait disorders muscle strengthening exercises relaxation exercises
Other: hippotherapy-assisted physiotherapy — The patients will be placed on the simulator and the starting position will be taught. your simulator before the application and in order to maintain the starting position throughout their movements.
  they will be warned during the applications.. Hippotherapy simulator is almost like walking.
  pattern and will be run in the 1st stage of the 3-stage speed level.
  Arms: hippotherapy group

SUMMARY:
The aim of the study is to examine the effect of hippotherapy simulator on trunk control, balance and gait in children with spastic diplegia cerebral palsy and its relationship with quality of life.

DETAILED DESCRIPTION:
Patients diagnosed with spastic diplegia cerebral palsy in the study; It will be classified according to Gross Motor Function Classification System (KMFSS). The Trunk Control Measurement Scale will be used to assess trunk control. Pediatric Berg Balance Scale will be used to assess balance. The 1 Minute Walk Test and the Timed Get Up and Go test will be used to assess walking. The WEEFIM scale will be used to assess quality of life. The study sample will be divided into two groups. The first group will receive 45 minutes of conventional physical therapy. In addition to 45 minutes of physical therapy, the other group will receive 15 minutes of hippotherapy simulator. The results will be compared at the beginning and end of the study.

Then, individuals will be divided into two groups with a simple randomized method. Traditional physical therapy will be applied to the control group for 45 minutes, 2 days a week, for 8 weeks. In addition to traditional physical therapy, 15 minutes of therapy training with a hippotherapy device will be applied to the experimental group. Evaluation tests will be repeated at the beginning and end of the study. Pre- and post-intervention data were statistically analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Diplegic Cerebral Palsy between the ages of 4 and 16
* Levels 1,2 and 3 according to KMFSS
* Have not had botox or surgery in the last 6 months
* Able to perceive simple commands
* Patients who can sit in the hippotherapy simulator will be included.

Exclusion Criteria:

* With hip dislocation
* Those with hearing or visual disabilities
* Those who do not want to be involved in the study
* Adductor spasticity is stage 3 and above according to the ashworth spasticity scale.
* With upper extremity amputation

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Pediatric Berg Balance Scale | 10 weeks
  Berg Balance Scale was designed for children to evaluate functions in activities of daily living.
  version. The scale consists of 14 assessments and each section is scored between 0-4; The highest possible score is 56.
Trunk Control Measurement Scale | 10 weeks
  For this reason, the scale consists of two parts: Static Sitting Balance (SSB) and Dynamic Sitting Balance (DSB). The DSB section also consists of two sub-parameters as selective motion control and dynamic reach. While the static sitting balance subscale evaluates static trunk control during lower and upper extremity movements, the selective motion control subscale evaluates selective trunk movements in three planes (flexion/extension, rotation, and lateral flexion). The dynamic reach subscale evaluates performance during reaching tasks that require active trunk movement. The scale consists of 15 items in total (subscales 5, 7 and 3 items, respectively). Items are scored on a 2, 3, and 4-point ordinal scale and are administered bilaterally when clinically significant. While the total score of the scale varies between 0-58 points, higher scores indicate a better performance.
1 Minute Walk Test | 10 weeks
  First, the child puts on his own clothes and shoes. He is allowed to use his splints and suitable walking aid. At least 5 minutes before starting the test. He is allowed to rest and then brought to the starting point of the path he will walk. When the command is given, it is said to start walking as fast as possible for 1 minute. It is also reported that he is not allowed to run. The distance is then calculated.
Timed get up and go test | 10 weeks
  It is a test used to measure mobility and assesses walking speed, postural control, functional mobility and balance. The Timed Get Up and Go Test measures the time it takes for a person to get up from an arm-supported chair, turn by walking 3 m, and walk back to the chair, then sit down. The time it takes to get up from the chair and sit back on the chair is recorded.
Functional independence measurement for children (WEEFIM) | 10 weeks
  It was developed to assess the level of functional independence of children with a physical disability and consists of three main categories and a total of 18 questions. A total of 18 questions under the heading of self-care, mobility and cognitive function categories are scored between 1 and 7. According to this; While performing the function to be evaluated, the child with a physical disability gets 1 point if he/she does it completely with assistance, and 7 points if he/she does it completely independently. The lowest score that the child can get from the scale is 18, and the highest score is 126.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin GÜNEŞ, Study Chair — Uskudar University
Locations (1):
- İşbir Hospital, Tuzla, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matusiak-Wieczorek E, Dziankowska-Zaborszczyk E, Synder M, Borowski A. The Influence of Hippotherapy on the Body Posture in a Sitting Position among Children with Cerebral Palsy. Int J Environ Res Public Health. 2020 Sep 19;17(18):6846. doi: 10.3390/ijerph17186846. PMID 32961681
- [Background] Hausler M, Heussen N. Protocol for a systematic review and meta-analysis on the effect of hippotherapy and related equine-assisted therapies on motor capabilities in children with cerebral palsy. Syst Rev. 2020 Mar 5;9(1):48. doi: 10.1186/s13643-020-01297-7. PMID 32138777
- [Background] Hyun C, Kim K, Lee S, Ko N, Lee IS, Koh SE. The Short-term Effects of Hippotherapy and Therapeutic Horseback Riding on Spasticity in Children With Cerebral Palsy: A Meta-analysis. Pediatr Phys Ther. 2022 Apr 1;34(2):172-178. doi: 10.1097/PEP.0000000000000880. PMID 35184078
- [Background] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598
- [Background] Apolo-Arenas MD, Jeronimo AFA, Cana-Pino A, Fernandes O, Alegrete J, Parraca JA. Standardized Outcomes Measures in Physical Therapy Practice for Treatment and Rehabilitation of Cerebral PALSY: A Systematic Review. J Pers Med. 2021 Jun 26;11(7):604. doi: 10.3390/jpm11070604. PMID 34206816